CLINICAL TRIAL: NCT00506012
Title: Phase II Efficacy and Safety of Taro Pharmaceuticals' Pro-Drug T2000 (1,3-Dimethoxymethyl-5,5-Diphenyl-Barbituric Acid) In Patients With Myoclonus Dystonia: An Open Label Sequential Dose Escalation Study
Brief Title: Pilot Efficacy Study of T2000 in Myoclonus Dystonia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow Recruitment of eligible patients
Sponsor: Sun Pharmaceutical Industries, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T2000-0633
Record Dates: First submitted 2007-07-20; First posted 2007-07-25 (Estimated); Last update posted 2013-12-23 (Estimated); Status verified 2013-11

CONDITIONS: Myoclonus
Keywords: Myoclonus Dystonia; Essential Myoclonus; Inherited Myoclonus; Dyskinesia; Movement Disorder
MeSH Terms: conditions — Myoclonus; Myoclonic dystonia; Dyskinesias; Movement Disorders

ARMS (1):
- 1 (Experimental): T2000
  Interventions: Drug: T2000

INTERVENTIONS:
Drug: T2000 — T2000 at doses of 200 mg a day to 1000 mg a day

SUMMARY:
This pilot study will evaluate the safety and efficacy of once daily T2000 when used to treat patients with Myoclonus Dystonia over a 12 week period.

DETAILED DESCRIPTION:
Myoclonus Dystonia (M-D) is a rare, inherited movement disorder in which patients experience myoclonus - sudden, brief, jerky involuntary motions, often in association with dystonia - involuntary sustained contractions causing twisting or abnormal posture. While most M-D patients respond significantly to alcohol, there are no approved medications for M-D. A variety of medications are currently used to treat M-D, but these treatments work in a small proportion of patients and provide only partial improvement in symptoms; their use is also limited by side-effects in many patients.

T2000 is a medication currently under development for the treatment of movement disorders, including essential tremor (ET). Although T2000 is a new medication, it belongs to a class of medications that has been used for many years for the treatment of a variety of medical conditions. In previous studies, T2000 appeared to be effective in controlling symptoms of ET and some patients with severe ET had major improvements in tremor. As would be expected for medications in this class, T2000 can cause sedation at high blood levels, such as may be seen when large doses are given to older individuals. In younger patients, T2000 caused only minimal side effects even when administered at high doses and for periods of several weeks to several months.

The current study will evaluate the safety and efficacy of T2000 in patients with M-D. Patients will receive doses of T2000 beginning at 200 mg a day and increasing every other week by an additional 200 mg a day up to a maximal dose of 1000 mg a day. The total duration of treatment will be 12 weeks. Patient's symptoms of myoclonus and dystonia, as well as overall neurological examination, will be monitored throughout the study. The response to T2000 will be determined by comparing the severity of myoclonus and dystonia while patients are receiving T2000 compared to the symptoms observed without active medication.

ELIGIBILITY:
Inclusion Criteria:

* Patients should meet diagnostic criteria for M-D based on the following criteria:

  * myoclonus is the primary feature; focal or segmental dystonia of any severity may also be present
  * symptoms began by age 20
  * a familial pattern should be present
  * neurological history should not be suggestive of a different neurological condition
  * investigations such as imaging, EEG and evoked potential tests should be normal
* Patients will be eligible for this study if they are symptomatic on their current treatment, cannot tolerate current therapies, or are treatment naïve patients who have been explained treatment alternatives.

Exclusion Criteria:

* Patients adequately controlled without side effects on a current M-D treatment
* Current treatment with a barbiturate such as phenobarbital or primidone
* Pregnant patients or patients who may become pregnant during the study
* Patients who must take medications that alter liver metabolism as well as patients with liver disease or coagulation disorders
* Patients with seizure disorders
* Patients with a history of allergy or hypersensitivity reaction to barbiturates or other related medications, such as phenobarbital or phenytoin
* Patient with significant general medical or clinical laboratory abnormalities

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2007-08; Primary Completion 2011-08 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Effect of treatment on the movement disorder will be measured by a myoclonus scale and a dystonia scale as well as by assessment of overall functional status. Response at various dosages will be compared to baseline for all patients. | Up to 12 weeks

SECONDARY OUTCOMES:
Safety parameters including neurological examination, blood tests and EKG will be monitored throughout the treatment period and during withdrawal of the medication. | Up to 16 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Investigator Site, Toronto, Ontario, Canada

REFERENCES:
- [Background] Melmed C, Moros D, Rutman H. Treatment of essential tremor with the barbiturate T2000 (1,3-dimethoxymethyl-5,5-diphenyl-barbituric acid). Mov Disord. 2007 Apr 15;22(5):723-7. doi: 10.1002/mds.21321. PMID 17265458